CLINICAL TRIAL: NCT06560814
Title: Non-surgical Interventions for Infertility in Endometriosis: A Parallel-Design Randomized Clinical Trial
Brief Title: Non-surgical Interventions for Infertility in Endometriosis
Acronym: RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Shakeela Ishrat, Associate Professor, Department of Reproductive Endocrinology & Infertility, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2021/06
Record Dates: First submitted 2021-03-11; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis; Infertility, Female
Keywords: endometriosis
MeSH Terms: conditions — Endometriosis; Infertility, Female | interventions — Cabergoline; Dydrogesterone; Progest

STUDY DESIGN:
Intervention Model Description: Open label, Parallel design randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabergoline (Experimental): Tab Cabergoline 0.5 mg twice weekly for 24 weeks, plus timed intercourse
  Interventions: Drug: Cabergoline plus timed intercourse
- Dydrogesterone (Active Comparator): tab Dydrogesterone( 10 mg) twice daily from day 5 to day 25 of menstrual cycle for 24 weeks, plus timed intercourse
  Interventions: Drug: Dydrogesterone plus timed intercourse

INTERVENTIONS:
Drug: Cabergoline plus timed intercourse — Cabergoline 0.5 mg tab orally twice weekly (fridays and tuesdays) after meal at night for 24 weeks plus intercourse timed with LH kit
  Other Names: Cabergol
  Arms: Cabergoline
Drug: Dydrogesterone plus timed intercourse — Dydrogesterone 10 mg tab orally twice daily from day 5 to day 25 of menstrual cycle for 24 weeks plus intercourse timed with LH kit
  Other Names: Progest
  Arms: Dydrogesterone

SUMMARY:
A parallel design randomized clinical trial was carried out on 18 women with clinically diagnosed endometriosis who wish pregnancy in the Department of Reproductive Endocrinology and Infertility, Bangabandhu Sheikh Mujib Medical University, (BSMMU), Shahbag, Dhaka. Those who voluntarily provide consent to participate in this study will be randomly allocated to one of the two treatment arms. Allocation concealment will be done by sequentially numbered sealed envelopes. The arms and interventions are cabergoline (0.5 mg twice weekly for 6 months, plus timed intercourse) and dydrogesteron (20 mg daily from day 5 to day 25 of menstrual cycle for 6 months, plus timed intercourse).The women will be assessed by telephone interview at monthly intervals, TVS and serum Ca 125 at 3 months and 6 months.

DETAILED DESCRIPTION:
Infertile women with endometriosis will be recruited from those attending Dept of Reproductive Endocrinology and Infertility after clinical diagnosis on the basis of sonographic findings of chocolate cyst with or without dysmenorrhea. After evaluating for eligibility criteria and taking informed consent she will be randomized to either cabergoline group or to dydrogesterone group. Women assigned to cabergoline group will receive 0.5 mg cabergoline twice weekly (fridays and tuesdays), after meal at night for 6 months. The dydrogesterone group will receive 10 mg of dydrogesterone twice daily from day 5 to day 25 of menstrual cycle for six months. She will be followed up every month to check for compliance or any side effects. The couple will have intercourse timed with LH kit or intercourse on alternate days from day 10 to day 15 of the cycle if the LH kit is not available. She will visit 3 months and 6 months after the beginning of treatment. At each follow up visit, she will be assessed for pregnancy, visual analog scale for pain and transvaginal sonogram to measure the chocolate cyst. Estimation of serum CA125 and any side effects will be noted.

ELIGIBILITY:
Inclusion Criteria:

1. Women of reproductive age 18-35 yrs
2. Women who are infertile or wish pregnancy
3. Sonographic diagnosis of chocolate cyst with or without dysmenorrhea
4. Women staying with her husband

Exclusion Criteria:

1. Recurrent endometrioma after previous surgery
2. BMI at or more than 30 kg/m2
3. Significant abnormalities in renal and liver function.
4. Known male factor
5. Use of investigational drugs or hormones, concomitant or in last 30 days.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 18 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain reduction estimated by mean change on a Visual Analog Scale | 24 weeks
  Mean change in Visual Analogue Score (1-10), higher score means worse outcome
Percentage change in size | 24 weeks
  Percentage change in size (maximum diameter) of chocolate cyst assessed by transvaginal ultrasound at week 24
Pregnancy rate | 24 weeks
  Proportion in each group of participants of those who conceive , biochemical (serum beta hCG > 40 IU/mL) or clinical (sonographic appearance of gestational sac)

SECONDARY OUTCOMES:
Change in CA 125 | 24 weeks
  Serum CA 125 level will be measured in blood
Adverse effect | 24 weeks
  From patient drug history

CONTACTS AND LOCATIONS:
Overall Officials: Shakeela Ishrat, FCPS Obgyn, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh